CLINICAL TRIAL: NCT02792777
Title: Concept Mapping as a Scalable Method for Identifying Patient-Important Outcomes
Acronym: VOICe
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 15G.667
Record Dates: First submitted 2016-06-02; First posted 2016-06-08 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Concept Mapping Versus Interviews
Keywords: Concept Mapping; VOICe; Interviews; Patient-Centered Research
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Interviews: Interview participants will be recruited from 3 different care settings: an acute care visit (in the emergency department), a post-acute care visit (within 1 week of a hospital discharge), and a routine primary care visit. Target sample size within each healthcare setting is 30 patients, which is the anticipated number needed for thematic saturation. The total recruitment goal for this cohort is 90-120 participants.
  Interventions: Other: Interviews
- Concept Mapping: Concept mapping participants will be recruited from existing clinical and research databases for 3 separate concept mapping groups, each with a target of 20 patients. The total recruitment goal for this cohort is 60 people.
  Interventions: Other: Concept Mapping (CM)

INTERVENTIONS:
Other: Interviews — Patients will be engaged in open-ended, semi-structured qualitative interviews, which will be performed one-on-one either in person or over the phone (depending on the healthcare setting that they are recruited from). Qualitative interviews will be audio recorded, with the patient's permission, transcribed, de-identified and entered into NVivo software for coding and analysis.
  Groups: Interviews
Other: Concept Mapping (CM) — The CM process consists of 3 steps that take place over 3 sessions:
  Step 1: Generation of Ideas- Participants brainstorm and generate responses to the focus statement. Once the group agrees that no new statements are being generated, the list of statements is reviewed within the group.
  Step 2: Structuring of Statements- Each participant is given a set of sort cards and asked to sort the statements into piles. Participants then rate each idea regarding importance. Research staff enters this information into the CM software.
  Concept Systems Global Software generates point maps using a technique that detects underlying similarities/differences between statements. The CM software then uses hierarchical cluster analysis to draw boundaries around the point map to create conceptual clusters.
  Step 3: Interpretation- The CM group revises the concept map. Participants review the cluster names suggested by the software and decide upon final naming of each cluster as a group.
  Groups: Concept Mapping

SUMMARY:
The goal of this study is to improve the methods with which researchers identify patient centered outcomes for use in research. Specifically, the investigators will test the application of concept mapping as compared to one-on-one interviews as a comprehensive and efficient method of identifying patient-important outcomes for use in research.

DETAILED DESCRIPTION:
This is an observational study comparing two methods - concept mapping and one-on-one interviews. The investigators will test the methods themselves by comparing the comprehensiveness of the lists of patient-important outcomes obtained through each method (primary outcome) as well as the efficiency, as measured by resource intensiveness, of the methods (secondary outcome). The aims of this study will be tested with adult patients with moderately to poorly controlled diabetes mellitus who receive care at a large, urban, academic health system. In order to allow comparisons of the comprehensiveness of the methods in producing patient-important outcomes regardless of the healthcare setting in which outcomes are elicited, the investigators will recruit patients for the interview group from 3 different care settings: an acute care visit (in the emergency department), a post-acute care visit (within 1 week of a hospital discharge), and a routine primary care visit. Target sample size within each healthcare setting is 30 patients, which is the anticipated number needed for thematic saturation. The investigators will then recruit patient-participants from existing clinical and research databases for 3 separate concept mapping groups, each with a target of 20 patients. In Aim 2, the investigators will test the hypothesis that concept mapping in a research setting produces outcomes consistent with those elicited from patients in the "real-world" settings. In Aim 3, the investigators will assess the overall resource utilization, assessed primarily by time required from patients, the research team, and the advisory board, of qualitative interviews conducted to thematic saturation within a single healthcare setting compared to resources used for a single iteration of concept mapping.

Findings from this work will improve patient-centered outcomes research methods by providing researchers with information about standardized scalable methods to identify patient-important outcomes for use in research studies, so that individual patients are able to select outcomes that are most useful to them. In addition to providing insight regarding methods for eliciting patient-centered outcomes, the study will also provide valuable information to stakeholders regarding how patients' priorities vary across the care continuum. The investigators will report how findings from concept mapping apply across healthcare settings, and the degree to which patient priorities (based on interviews) differ across healthcare settings. If concept mapping results (collected in the research setting) capture the priorities identified by patients across different healthcare settings, this finding would enhance researchers' ability to perform studies in different, or multiple, settings. If the findings do not generalize across settings, this will be a valuable finding demonstrating that patient priorities differ across interview settings and patient acuity and will validate researchers' needs to be specific about the setting in which they choose to perform research to ensure they are reaching their intended patient population.

The work is being performed in close collaboration with the Patient and Key Stakeholder Advisory Board (PAKSAB) - equal partners with the research team who have been involved with the proposal from inception. PAKSAB members will be part of the research team throughout conducting the aims and assisting with all analysis and data interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age 18 and older)

  * English speaking
  * Provide informed consent
* Diagnosis of moderately to poorly controlled diabetes mellitus (DM) defined as follows (for interview groups):

  * Acute care setting: patient in the Jefferson Emergency Department (ED) for a diabetes-related problem determined to require medical treatment
  * Post-acute care setting: patient was discharged from the Jefferson Family Medicine Associates (JFMA) hospital service within the past 7 days after admission for a diabetes-related problem
  * Primary care setting: patient currently attending a routine scheduled care visit (not urgent need) at the JFMA practice and has at least 2 measurements of HgbA1C > 7.5 in the prior one year
* Diagnosis of moderately to poorly controlled diabetes mellitus (DM) defined as follows (for concept mapping groups):

  * Acute care setting: patient within the Jefferson ED patient contact database (see below) who has had a visit to the Jefferson ED over the past 6 months (as determined on chart review) for a diabetes-related problem
  * Post-acute care setting: patient was discharged from the JFMA hospital service within the past 6 months after admission for a diabetes-related problem
  * Primary care setting: patient has had routine scheduled office visit within the past 6 months to the JFMA practice and has at least 2 measurements of HgbA1C > 7.5 in the prior one year

Exclusion Criteria:

* Patient has had a significant permanent complication related to DM including:

  * End stage renal disease
  * History of amputation
  * Blindness related to diabetes complication
* Patient undergoing medical clearance for a detox center or any involuntary court or magistrate order
* Patient in police custody or currently incarcerated individual
* Patient who has, in their clinician's best judgment, major communication barriers such as visual or hearing impairment or dementia that would compromise their ability to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators aim to engage a discrete population of patients who have recently sought care at Thomas Jefferson University for treatment needs related to moderately to poorly controlled diabetes. Consistent with the overall population served by Jefferson, the investigators expect greater than 50% of enrolled patients to be African American and approximately 30% of them to be at the <20% federal poverty line. All data will be collected prospectively. The investigators decided to engage patients with moderately to poorly controlled DM because these patients have a known high risk of severe complications related to poor diabetes control, and a significant proportion of patients remain poorly controlled despite available therapies. The investigators thus determined in discussion with the PAKSAB that this population is a good candidate for testing the method of concept mapping to identify patient-important outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01-29 (Actual); Study Completion 2018-03-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ThomasJeffersonU, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gentsch AT, Reed MK, Cunningham A, Chang AM, Kahn S, Kovalsky D, Doty AMB, Mills G, Hollander JE, Rising KL. "Once I take that one bite": the consideration of harm reduction as a strategy to support dietary change for patients with diabetes. BMC Endocr Disord. 2024 Jan 2;24(1):3. doi: 10.1186/s12902-023-01529-6. PMID 38166864
- [Derived] LaNoue M, Gentsch A, Cunningham A, Mills G, Doty AMB, Hollander JE, Carr BG, Loebell L, Weingarten G, Rising KL. Eliciting patient-important outcomes through group brainstorming: when is saturation reached? J Patient Rep Outcomes. 2019 Feb 4;3(1):9. doi: 10.1186/s41687-019-0097-2. PMID 30714080
- [Derived] Rising KL, LaNoue M, Gentsch AT, Doty AMB, Cunningham A, Carr BG, Hollander JE, Latimer L, Loebell L, Weingarten G, White N, Mills G. The power of the group: comparison of interviews and group concept mapping for identifying patient-important outcomes of care. BMC Med Res Methodol. 2019 Jan 8;19(1):7. doi: 10.1186/s12874-018-0656-x. PMID 30621586

RESULTS

PARTICIPANT FLOW:
Groups:
- Concept Mapping: Concept mapping participants will be recruited from existing clinical and research databases for 3 separate concept mapping groups, each with a target recruitment of 20 patients. The total recruitment goal for this cohort is 60 people.
  Concept Mapping (CM): The CM process consists of 3 steps that take place over 3 sessions:
  Step 1: Generation of Ideas- Participants brainstorm responses to a focus statement.
  Step 2: Structuring of Statements- Each participant is given a set of sort cards and asked to sort the statements into piles. Participants then rate each idea regarding importance.
  CM Software detects underlying similarities/differences between statements to generate point maps. The CM software then uses hierarchical cluster analysis to draw boundaries around the point map to create conceptual clusters.
  Step 3: Interpretation- The CM group revises the concept map. Participants review cluster names suggested by the software and decide upon final naming of each cluster.
Period: Overall Study
Arm/Group | Interviews | Concept Mapping
Started | 96 | 52
Completed | 89 | 52
Not Completed | 7 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Recording malfunction | 2 | 0
Not completed — Later determined to be ineligible | 2 | 0
Not completed — Participant interviewed twice | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interviews | Concept Mapping | Total
Number analyzed (Participants) | 89 | 52 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (13.8) | 55.6 (14.7) | 54.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant declined to answer, did not collect data from 1 participant
  Participants
    number analyzed (Participants) | 89 | 50 | 139
    Female | 49 | 24 | 73
    Male | 40 | 26 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 80 | 49 | 129
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 60 | 42 | 102
  Race: Caucasian/White | 24 | 5 | 29
  Race: Other | 4 | 4 | 8
  Race: Unknown or not reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 89 | 52 | 141

OUTCOME MEASURES:

1. Primary Outcome: Comprehensiveness of Interviews as Compared to One Concept Mapping Group
Description: The investigators will use a qualitative content analysis approach to analyze interview transcripts from one healthcare setting, with one of the codes being "goals". All ideas coded to "goals" that are in any way relevant to patients' diabetes care will be extracted to create a list of patient-important outcomes. The investigators will then determine the proportion of patient-important outcomes identified in the interviews from one healthcare setting that are present in the list of patient-important outcomes generated from the initial concept mapping group during the brainstorming session. The investigators will also identify the presence of unique outcomes found in each method.
Time Frame: Interviewed patients participated for 1 day; Concept mapping patients participated for 3 days
Measure: Number; unit: Reported patient-important outcomes
Arm/Group | Interviews | Concept Mapping
Number analyzed (Participants) | 30 | 24
Reported patient-important outcomes
  Total number of outcomes | 26 | 33
  Number of unique outcomes | 6 | 13

2. Primary Outcome: Comprehensiveness of Interviews Compared to Three Concept Mapping Groups
Description: The investigators will use a qualitative content analysis approach to analyze interview transcripts, with one of the codes being "goals". All ideas coded to "goals" that are in any way relevant to patients' diabetes care will be extracted to create a list of patient-important outcomes. The investigators will then determine the proportion of patient-important outcomes identified in interviews that are present in an aggregate list of patient-important outcomes generated from the brainstorming session of all three concept mapping groups. The investigators will also identify the presence of additional patient-important outcomes in three concept mapping groups that were not identified in interviews.
Time Frame: Interviewed patients participated for 1 day; One group of concept mapping patients participated for 3 days
Measure: Number; unit: Reported patient-important outcomes
Arm/Group | Interviews | Concept Mapping
Number analyzed (Participants) | 89 | 52
Reported patient-important outcomes
  Total Number of Outcomes | 26 | 38
  Unique Number of Outcomes | 3 | 15

3. Primary Outcome: Comprehensiveness of Concept Mapping
Description: The investigators will measure the comprehensiveness of outcomes elicited in one concept mapping group compared to multiple groups. The investigators will assess "concept mapping saturation," wherein we compare the patient-important outcomes that emerge from each CM group. The investigators will use the outcomes from our first group as the "baseline data," and will determine the amount of new data added from including a second/third group. This assessment will allow us to draw a basic "concept mapping saturation curve."
Time Frame: 3 days for one concept mapping group
Population: This analysis is of the number of patient-important outcomes per concept mapping group.
Measure: Number; unit: Reported patient-important outcomes
Arm/Group | Concept Mapping
Number analyzed (Participants) | 52
Reported patient-important outcomes
  One Group: number analyzed (Participants) | 24
  One Group | 33
  Two Groups: number analyzed (Participants) | 14
  Two Groups | 36
  Three Groups: number analyzed (Participants) | 14
  Three Groups | 38

4. Secondary Outcome: Comparison of Method Efficiency in Terms of Time
Description: The investigators will assess the efficiency of implementation of the two methods, with efficiency including time required by researchers (team of 3) and patient-participants to complete each method. The investigators will compare the efficiency of conducting one concept mapping iteration (24 participants) to the efficiency of performing one set of interviews done to theme saturation (30 interviews). This efficiency analysis is structured for what would need to be budgeted in a grant application, and will provide useful information for general planning needs for method implementation.
Time Frame: Interviewed patients participated for 1 day; Concept mapping patients participated for 3 days
Measure: Number; unit: Hours
Arm/Group | Interviews | Concept Mapping
Number analyzed (Participants) | 30 | 24
Hours
  Patient travel | 0 | 2
  Patient participation | 1 | 6
  Research team trainings | 20 | 11
  Research team participant recruitment | 66 | 59
  Research team travel | 60 | 12
  Research team conducting method | 38 | 18
  Research team data analysis | 133 | 4

5. Secondary Outcome: Comparison of Method Efficiency in Terms of Cost
Description: The investigators will assess the efficiency of implementation of the two methods, with efficiency assessed by cost to complete a single concept mapping iteration (24 participants) and cost to complete one set of interviews performed to saturation (30 interviews). This efficiency analysis is structured for what would need to be budgeted in a grant application, and will provide useful information for general planning needs for method implementation.
Time Frame: Interviewed patients participated for 1 day; Concept mapping patients participated for 3 days
Measure: Number; unit: Dollars
Arm/Group | Interviews | Concept Mapping
Number analyzed (Participants) | 30 | 24
Dollars
  Patient Incentives | 750 | 3,000
  Transcription | 1,000 | 0
  Data Analysis Software | 1,380 | 2,000

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Description: All-Cause Mortality, Serious, and Other [not including Serious] Adverse Events were not monitored or assessed because patients were not at risk for adverse events aside from discomfort during interviews and concept mapping sessions.
Arm/Group | Interviews | Concept Mapping
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Limited generalizability due to all enrollments in same health system; Potential selection bias to more engaged/motivated patients; Method efficiency may vary depending on size of research team, patient incentives, and analysis software needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT02792777/Prot_SAP_000.pdf